CLINICAL TRIAL: NCT03227393
Title: The Effect of Yoga on Cardiac Sympathetic Innervation Evaluated by I-123 mIBG
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was not opened at site.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Mehran Attari, Professor of Medicine, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015-7643
Record Dates: First submitted 2017-07-20; First posted 2017-07-24 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure, Systolic
Keywords: Heart Failure, Systolic; Defibrillators, Implantable; Pacemaker, Artificial
MeSH Terms: conditions — Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No yoga training (No Intervention): This will be the control arm. The patients in this arm will not receive any yoga training. They will be continued on all their home, guideline-directed heart failure medications. They will undergo the same baseline and study completion evaluation as the treatment arm, including an I-123 MIBG scan, 24-hour holter monitoring and device interrogation.
- Yoga training (Experimental): The patients in this arm will receive yoga training. This includes weekly group yoga sessions consisting of breathing exercises, yoga poses, and relaxation and meditation lasting for about 80-90 minutes total. Patients will be asked to do home yoga practices at least twice a week and to document the date and time. Patients in this arm will have the same baseline and study completion evaluation as the control arm, including an I-123 MIBG scan, 24-hour holter monitoring and device interrogation.
  Interventions: Behavioral: Yoga training

INTERVENTIONS:
Behavioral: Yoga training — Subjects will complete in class yoga training weekly for 8 weeks with additional practice at home
  Arms: Yoga training

SUMMARY:
The purpose of this study is to evaluate if yoga practice will reduce cardiac sympathetic activity and subsequently cardiac arrhythmias.

DETAILED DESCRIPTION:
Subjects with reduced ejection fraction will be randomized to 8 weeks Yoga training (1 in class session and home practice) vs. no Yoga. They will undergo holter monitoring, cardiac device interrogation, and I-123 mIBG imaging at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test in females
* Ejection Fraction </= 40% assessed by echocardiogram within the last 12 months
* Stable dose of heart failure medications including afterload reducing medication such as ACE-I, ARB and hydralazine; beta blockers; digoxin and aldosterone antagonist for at least 4 months and no anticipated changes for 8 weeks. (i.e. no greater than a 50% dose change within the past month)
* Has an implantable pacemaker or ICD
* NYHA II-IV

Exclusion Criteria:

* pregnant or lactating female
* females without a pregnancy test
* co-administration of a positive inotrope (i.e. milrinone or dobutamine)
* history of significant medical non-compliance
* unwilling to adhere to the protocol
* Orthopedic limitation making yoga participation difficult
* Underlying cardiac rhythm other than sinus rhythm
* Recent history within 6 months prior to enrollment of unstable coronary artery disease (unstable angina, recent heart attack, recent revascularization, or decompensated heart failure)
* implantation of a cardiac resynchronization therapy device in the past 3 months.
* TIA, CVA, or major surgery in the past 3 months
* iodine or adreview (123-MIBG) allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Cardiac sympathetic activity following yoga training | 8 weeks
  A comparison of of the I-123 MIBG heart to mediastinal uptake ratio at baseline and completion of the yoga training.

SECONDARY OUTCOMES:
Relationship between I-123MIBG heart-to-mediastinal ratios and the total atrial and ventricular arrhythmia burden. | 8 weeks
  Association between heart to mediastinum ration and ventricular arrhythmia burden

CONTACTS AND LOCATIONS:
Overall Officials: Mehran Attari, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Thrall G, Lip GY, Carroll D, Lane D. Depression, anxiety, and quality of life in patients with atrial fibrillation. Chest. 2007 Oct;132(4):1259-64. doi: 10.1378/chest.07-0036. Epub 2007 Jul 23. PMID 17646231
- [Background] Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Kay GN, Le Huezey JY, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann LS. 2011 ACCF/AHA/HRS focused updates incorporated into the ACC/AHA/ESC 2006 Guidelines for the management of patients with atrial fibrillation: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines developed in partnership with the European Society of Cardiology and in collaboration with the European Heart Rhythm Association and the Heart Rhythm Society. J Am Coll Cardiol. 2011 Mar 15;57(11):e101-98. doi: 10.1016/j.jacc.2010.09.013. No abstract available. PMID 21392637
- [Background] Cheriyath P, He F, Peters I, Li X, Alagona P Jr, Wu C, Pu M, Cascio WE, Liao D. Relation of atrial and/or ventricular premature complexes on a two-minute rhythm strip to the risk of sudden cardiac death (the Atherosclerosis Risk in Communities [ARIC] study). Am J Cardiol. 2011 Jan 15;107(2):151-5. doi: 10.1016/j.amjcard.2010.09.002. PMID 21211594
- [Background] Florea VG, Cohn JN. The autonomic nervous system and heart failure. Circ Res. 2014 May 23;114(11):1815-26. doi: 10.1161/CIRCRESAHA.114.302589. PMID 24855204
- [Background] La Rovere MT, Pinna GD, Hohnloser SH, Marcus FI, Mortara A, Nohara R, Bigger JT Jr, Camm AJ, Schwartz PJ; ATRAMI Investigators. Autonomic Tone and Reflexes After Myocardial Infarcton. Baroreflex sensitivity and heart rate variability in the identification of patients at risk for life-threatening arrhythmias: implications for clinical trials. Circulation. 2001 Apr 24;103(16):2072-7. doi: 10.1161/01.cir.103.16.2072. PMID 11319197
- [Background] La Rovere MT, Pinna GD, Maestri R, Mortara A, Capomolla S, Febo O, Ferrari R, Franchini M, Gnemmi M, Opasich C, Riccardi PG, Traversi E, Cobelli F. Short-term heart rate variability strongly predicts sudden cardiac death in chronic heart failure patients. Circulation. 2003 Feb 4;107(4):565-70. doi: 10.1161/01.cir.0000047275.25795.17. PMID 12566367
- [Background] Mitrani RD, Klein LS, Miles WM, Hackett FK, Burt RW, Wellman HN, Zipes DP. Regional cardiac sympathetic denervation in patients with ventricular tachycardia in the absence of coronary artery disease. J Am Coll Cardiol. 1993 Nov 1;22(5):1344-53. doi: 10.1016/0735-1097(93)90541-8. PMID 8227790
- [Background] Paul M, Schafers M, Kies P, Acil T, Schafers K, Breithardt G, Schober O, Wichter T. Impact of sympathetic innervation on recurrent life-threatening arrhythmias in the follow-up of patients with idiopathic ventricular fibrillation. Eur J Nucl Med Mol Imaging. 2006 Aug;33(8):866-70. doi: 10.1007/s00259-005-0061-7. Epub 2006 Apr 13. PMID 16612587
- [Background] Patterson E, Po SS, Scherlag BJ, Lazzara R. Triggered firing in pulmonary veins initiated by in vitro autonomic nerve stimulation. Heart Rhythm. 2005 Jun;2(6):624-31. doi: 10.1016/j.hrthm.2005.02.012. PMID 15922271
- [Background] Coccagna G, Capucci A, Bauleo S, Boriani G, Santarelli A. Paroxysmal atrial fibrillation in sleep. Sleep. 1997 Jun;20(6):396-8. doi: 10.1093/sleep/20.6.396. PMID 9302722
- [Background] Po SS, Yu L, Scherlag BJ. Cardiac autonomic nervous system: a tug of war between the big brain and little brain--friends or foes? Heart Rhythm. 2009 Dec;6(12):1780-1. doi: 10.1016/j.hrthm.2009.09.006. Epub 2009 Sep 6. No abstract available. PMID 19959129
- [Background] Shen MJ, Shinohara T, Park HW, Frick K, Ice DS, Choi EK, Han S, Maruyama M, Sharma R, Shen C, Fishbein MC, Chen LS, Lopshire JC, Zipes DP, Lin SF, Chen PS. Continuous low-level vagus nerve stimulation reduces stellate ganglion nerve activity and paroxysmal atrial tachyarrhythmias in ambulatory canines. Circulation. 2011 May 24;123(20):2204-12. doi: 10.1161/CIRCULATIONAHA.111.018028. Epub 2011 May 9. PMID 21555706
- [Background] Collura CA, Johnson JN, Moir C, Ackerman MJ. Left cardiac sympathetic denervation for the treatment of long QT syndrome and catecholaminergic polymorphic ventricular tachycardia using video-assisted thoracic surgery. Heart Rhythm. 2009 Jun;6(6):752-9. doi: 10.1016/j.hrthm.2009.03.024. Epub 2009 Mar 19. PMID 19467503
- [Background] Schwartz PJ, Priori SG, Cerrone M, Spazzolini C, Odero A, Napolitano C, Bloise R, De Ferrari GM, Klersy C, Moss AJ, Zareba W, Robinson JL, Hall WJ, Brink PA, Toivonen L, Epstein AE, Li C, Hu D. Left cardiac sympathetic denervation in the management of high-risk patients affected by the long-QT syndrome. Circulation. 2004 Apr 20;109(15):1826-33. doi: 10.1161/01.CIR.0000125523.14403.1E. Epub 2004 Mar 29. PMID 15051644
- [Background] Wilde AA, Bhuiyan ZA, Crotti L, Facchini M, De Ferrari GM, Paul T, Ferrandi C, Koolbergen DR, Odero A, Schwartz PJ. Left cardiac sympathetic denervation for catecholaminergic polymorphic ventricular tachycardia. N Engl J Med. 2008 May 8;358(19):2024-9. doi: 10.1056/NEJMoa0708006. PMID 18463378
- [Background] Bourke T, Vaseghi M, Michowitz Y, Sankhla V, Shah M, Swapna N, Boyle NG, Mahajan A, Narasimhan C, Lokhandwala Y, Shivkumar K. Neuraxial modulation for refractory ventricular arrhythmias: value of thoracic epidural anesthesia and surgical left cardiac sympathetic denervation. Circulation. 2010 Jun 1;121(21):2255-62. doi: 10.1161/CIRCULATIONAHA.109.929703. Epub 2010 May 17. PMID 20479150
- [Background] Thayer JF, Lane RD. The role of vagal function in the risk for cardiovascular disease and mortality. Biol Psychol. 2007 Feb;74(2):224-42. doi: 10.1016/j.biopsycho.2005.11.013. Epub 2006 Dec 19. PMID 17182165
- [Background] Desai MY, Watanabe MA, Laddu AA, Hauptman PJ. Pharmacologic modulation of parasympathetic activity in heart failure. Heart Fail Rev. 2011 Mar;16(2):179-93. doi: 10.1007/s10741-010-9195-1. PMID 20924667
- [Background] Pullen PR, Nagamia SH, Mehta PK, Thompson WR, Benardot D, Hammoud R, Parrott JM, Sola S, Khan BV. Effects of yoga on inflammation and exercise capacity in patients with chronic heart failure. J Card Fail. 2008 Jun;14(5):407-13. doi: 10.1016/j.cardfail.2007.12.007. Epub 2008 May 27. PMID 18514933
- [Background] Cramer H, Lauche R, Haller H, Dobos G, Michalsen A. A systematic review of yoga for heart disease. Eur J Prev Cardiol. 2015 Mar;22(3):284-95. doi: 10.1177/2047487314523132. Epub 2014 Feb 3. PMID 24491402
- [Background] Krishna BH, Pal P, G K P, J B, E J, Y S, M G S, G S G. Effect of yoga therapy on heart rate, blood pressure and cardiac autonomic function in heart failure. J Clin Diagn Res. 2014 Jan;8(1):14-6. doi: 10.7860/JCDR/2014/7844.3983. Epub 2014 Jan 12. PMID 24596712
- [Background] Krishna BH, Pal P, Pal G, Balachander J, Jayasettiaseelon E, Sreekanth Y, Sridhar M, Gaur G. A Randomized Controlled Trial to Study the Effect of Yoga Therapy on Cardiac Function and N Terminal Pro BNP in Heart Failure. Integr Med Insights. 2014 Apr 1;9:1-6. doi: 10.4137/IMI.S13939. eCollection 2014. PMID 24737932
- [Background] Pullen PR, Thompson WR, Benardot D, Brandon LJ, Mehta PK, Rifai L, Vadnais DS, Parrott JM, Khan BV. Benefits of yoga for African American heart failure patients. Med Sci Sports Exerc. 2010 Apr;42(4):651-7. doi: 10.1249/MSS.0b013e3181bf24c4. PMID 19952833
- [Background] Howie-Esquivel J, Lee J, Collier G, Mehling W, Fleischmann K. Yoga in heart failure patients: a pilot study. J Card Fail. 2010 Sep;16(9):742-9. doi: 10.1016/j.cardfail.2010.04.011. Epub 2010 Jun 8. PMID 20797598
- [Background] Vempati RP, Telles S. Yoga-based guided relaxation reduces sympathetic activity judged from baseline levels. Psychol Rep. 2002 Apr;90(2):487-94. doi: 10.2466/pr0.2002.90.2.487. PMID 12061588
- [Background] Khattab K, Khattab AA, Ortak J, Richardt G, Bonnemeier H. Iyengar yoga increases cardiac parasympathetic nervous modulation among healthy yoga practitioners. Evid Based Complement Alternat Med. 2007 Dec;4(4):511-7. doi: 10.1093/ecam/nem087. PMID 18227919
- [Background] Santaella DF, Devesa CR, Rojo MR, Amato MB, Drager LF, Casali KR, Montano N, Lorenzi-Filho G. Yoga respiratory training improves respiratory function and cardiac sympathovagal balance in elderly subjects: a randomised controlled trial. BMJ Open. 2011 May 24;1(1):e000085. doi: 10.1136/bmjopen-2011-000085. PMID 22021757
- [Background] Lakkireddy D, Atkins D, Pillarisetti J, Ryschon K, Bommana S, Drisko J, Vanga S, Dawn B. Effect of yoga on arrhythmia burden, anxiety, depression, and quality of life in paroxysmal atrial fibrillation: the YOGA My Heart Study. J Am Coll Cardiol. 2013 Mar 19;61(11):1177-82. doi: 10.1016/j.jacc.2012.11.060. Epub 2013 Jan 30. PMID 23375926
- [Background] Kiecolt-Glaser JK, Christian LM, Andridge R, Hwang BS, Malarkey WB, Belury MA, Emery CF, Glaser R. Adiponectin, leptin, and yoga practice. Physiol Behav. 2012 Dec 5;107(5):809-13. doi: 10.1016/j.physbeh.2012.01.016. Epub 2012 Jan 27. PMID 22306535
- [Background] Toise SC, Sears SF, Schoenfeld MH, Blitzer ML, Marieb MA, Drury JH, Slade MD, Donohue TJ. Psychosocial and cardiac outcomes of yoga for ICD patients: a randomized clinical control trial. Pacing Clin Electrophysiol. 2014 Jan;37(1):48-62. doi: 10.1111/pace.12252. Epub 2013 Aug 26. PMID 23981048
- [Background] Jacobson AF, Lombard J, Banerjee G, Camici PG. 123I-mIBG scintigraphy to predict risk for adverse cardiac outcomes in heart failure patients: design of two prospective multicenter international trials. J Nucl Cardiol. 2009 Jan-Feb;16(1):113-21. doi: 10.1007/s12350-008-9008-2. Epub 2009 Jan 20. PMID 19152136
- [Background] Jacobson AF, Senior R, Cerqueira MD, Wong ND, Thomas GS, Lopez VA, Agostini D, Weiland F, Chandna H, Narula J; ADMIRE-HF Investigators. Myocardial iodine-123 meta-iodobenzylguanidine imaging and cardiac events in heart failure. Results of the prospective ADMIRE-HF (AdreView Myocardial Imaging for Risk Evaluation in Heart Failure) study. J Am Coll Cardiol. 2010 May 18;55(20):2212-21. doi: 10.1016/j.jacc.2010.01.014. Epub 2010 Feb 25. PMID 20188504
- [Background] Narula J, Gerson M, Thomas GS, Cerqueira MD, Jacobson AF. (1)(2)(3)I-MIBG Imaging for Prediction of Mortality and Potentially Fatal Events in Heart Failure: The ADMIRE-HFX Study. J Nucl Med. 2015 Jul;56(7):1011-8. doi: 10.2967/jnumed.115.156406. Epub 2015 Jun 11. PMID 26069309
- [Background] Verschure DO, Veltman CE, Manrique A, Somsen GA, Koutelou M, Katsikis A, Agostini D, Gerson MC, van Eck-Smit BL, Scholte AJ, Jacobson AF, Verberne HJ. For what endpoint does myocardial 123I-MIBG scintigraphy have the greatest prognostic value in patients with chronic heart failure? Results of a pooled individual patient data meta-analysis. Eur Heart J Cardiovasc Imaging. 2014 Sep;15(9):996-1003. doi: 10.1093/ehjci/jeu044. Epub 2014 Mar 30. PMID 24686260
- [Background] Gerson MC, McGuire N, Wagoner LE. Sympathetic nervous system function as measured by I-123 metaiodobenzylguanidine predicts transplant-free survival in heart failure patients with idiopathic dilated cardiomyopathy. J Card Fail. 2003 Oct;9(5):384-91. doi: 10.1054/s1071-9164(03)00134-9. PMID 14583900
- [Background] Waqar F, Dunlap SH, Gerson MC. What will be the role of I-123 MIBG in improving the outcome of medically treated heart failure patients? J Nucl Cardiol. 2012 Dec;19(6):1198-205; quiz 1206-10. doi: 10.1007/s12350-012-9612-z. No abstract available. PMID 22956185
- [Background] Gerson MC, Dwivedi AK, Abdallah M, Shukla R, Jacobson AF. Significance of I-123 metaiodobenzylguanidine ((1)(2)(3)I-MIBG) lung activity in subjects with heart failure in comparison to healthy control subjects. J Nucl Cardiol. 2013 Aug;20(4):592-9. doi: 10.1007/s12350-013-9714-2. Epub 2013 Apr 30. PMID 23636966
- [Background] Gerson MC, Caldwell JH, Ananthasubramaniam K, Clements IP, Henzlova MJ, Amanullah A, Jacobson AF. Influence of diabetes mellitus on prognostic utility of imaging of myocardial sympathetic innervation in heart failure patients. Circ Cardiovasc Imaging. 2011 Mar;4(2):87-93. doi: 10.1161/CIRCIMAGING.110.954784. Epub 2010 Dec 30. PMID 21193691
- [Background] Mushtaq N, Gerson MC. I-123 metaiodobenzylguanidine imaging in non-insulin-dependent diabetic patients with normal myocardial perfusion scans: new insights into their increased cardiac morbidity and mortality rates. J Nucl Cardiol. 2006 Jan-Feb;13(1):8-10. doi: 10.1016/j.nuclcard.2005.11.005. No abstract available. PMID 16464711
- [Background] Gerson MC, Wagoner LE, McGuire N, Liggett SB. Activity of the uptake-1 norepinephrine transporter as measured by I-123 MIBG in heart failure patients with a loss-of-function polymorphism of the presynaptic alpha2C-adrenergic receptor. J Nucl Cardiol. 2003 Nov-Dec;10(6):583-9. doi: 10.1016/j.nuclcard.2003.07.001. PMID 14668769
- [Background] Gerson MC, Craft LL, McGuire N, Suresh DP, Abraham WT, Wagoner LE. Carvedilol improves left ventricular function in heart failure patients with idiopathic dilated cardiomyopathy and a wide range of sympathetic nervous system function as measured by iodine 123 metaiodobenzylguanidine. J Nucl Cardiol. 2002 Nov-Dec;9(6):608-15. doi: 10.1067/mnc.2002.127717. PMID 12466785
- [Background] Abdallah M, Gerson MC. A step forward in the use of SPECT imaging with I-123 MIBG. J Nucl Cardiol. 2012 Feb;19(1):16-8. doi: 10.1007/s12350-011-9495-4. No abstract available. PMID 22203444
- [Result] Kubo A, Hung YY, Ritterman J. Yoga for heart failure patients: a feasibility pilot study with a multiethnic population. Int J Yoga Therap. 2011;(21):77-83. PMID 22398347
- [Result] Barclay S, Momen N, Case-Upton S, Kuhn I, Smith E. End-of-life care conversations with heart failure patients: a systematic literature review and narrative synthesis. Br J Gen Pract. 2011 Jan;61(582):e49-62. doi: 10.3399/bjgp11X549018. PMID 21401993
- [Result] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990